CLINICAL TRIAL: NCT05652400
Title: HIV Transmission in the Era of Scaling up Access to Antiretroviral Therapy in Ethiopia
Brief Title: HIV Transmission in the Era of Scaling up Antiretroviral Therapy in Ethiopia
Acronym: THESA
Status: Active, not recruiting | Type: Observational
Sponsor: Lund University (Other)
Collaborators: Armauer Hansen Research Institute, Ethiopia (Other); Ethiopian Public Health Institute (Other Government); Oromia Regional Health Bureau (Unknown)
Responsible Party: Sponsor
Other Study IDs: LundU 2019-02627
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: HIV-1-infection; Antiretroviral Therapy
Keywords: HIV infection; Transmission; Drug resistance; Treatment monitoring; Ethiopia
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be collected from participants at inclusion and longitudinally during follow-up (2 years). Both plasma and whole blood samples will be stored at -80 C using individual codes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Individuals diagnosed with HIV infection: People with HIV
  Interventions: Other: Exposure to antiretroviral therapy

INTERVENTIONS:
Other: Exposure to antiretroviral therapy — Outcomes will be compared with regard to current or previous exposure to antiretroviral therapy.

SUMMARY:
The goal of this observational study is to understand patterns of HIV transmission in a high-prevalence area in Ethiopia, and to compare viral genetic information in people with HIV who are newly diagnosed and have not been exposed to antiretroviral therapy with persons receiving antiretroviral therapy without viral suppression.

The main questions it aims to answer are:

* Do people with HIV who fail to achieve viral suppression contribute to the ongoing spread of HIV in Ethiopia, or does HIV transmission mainly occur between persons with no exposure to such therapy?
* Are viruses with drug-resistance mutations transmitted onwards from people with HIV receiving antiretroviral therapy who fail to achieve viral suppression? * Which factors are involved in treatment failure and emergence of drug-resistant viruses longitudinally?

Participants will be enrolled with regard to history of antiretroviral therapy exposure (newly diagnosed/treatment-naïve vs. treatment-experienced with lack of viral suppression), using persons on antiretroviral therapy with viral suppression for control. We will compare the following outcomes between these groups:

* Clustering of viral genetic sequences at inclusion (implying linked transmission)
* Prevalence of drug-resistance-associated mutations at inclusion
* Viral suppression and emergence of drug-resistance mutations during follow-up

DETAILED DESCRIPTION:
Background Persons with incomplete viral suppression during antiretroviral therapy (ART) may harbor drug-resistant viruses, which have capacity for onwards transmission. The investigators hypothesize that individuals with previous or current exposure to ART contribute to HIV transmission, and that this includes transmission of drug-resistant viruses. This hypothesis is addressed by the use of molecular epidemiological analysis of viral sequences from persons newly diagnosed with HIV and those with ongoing viral replication during ART, combined with data on transmission risk behavior. In addition, based on findings described above, the investigators will include data on socio-demographic conditions in this analysis.

The chance of achieving viral suppression after treatment modification for persons with detectable viremia during ART is frequently compromised by the presence of drug-resistance mutations, adherence problems or irregular drug supply. There is limited data on the efficacy of dolutegravir (currently recommended as part of 1st and 2nd line ART regimens in sub-Saharan Africa) as a component of ART regimens in low-income settings. The investigators hypothesize that persons with incomplete viral suppression during prior ART are at increased risk of emergence of drug-resistance mutations during dolutegravir-based treatment, including mutations conferring dolutegravir resistance. The investigators will explore this hypothesis with deep sequencing of HIV RNA detected during longitudinal follow-up, with special regard to previous ART experience.

Methods Participants will be recruited and followed at public health facilities (hospitals and health centers) in the city of Adama and the surrounding area (population >600 000 inhabitants), located along the main transport highway in Ethiopia. The HIV prevalence in this area is considerably higher than the national average (9.3% among pregnant women).

Two categories of HIV-positive men and women aged >16 years are eligible for inclusion if specific criteria for the different categories (explained below) are met and written informed consent is provided.

i. Newly diagnosed persons; recruited in connection to HIV testing and/or first presentation to care, with no current or prior exposure to ART.

ii. Patients with current or prior exposure to ART; identified and recruited at ART clinics. In these clinics, all ART recipients are tested annually for viral load (VL; according to national guidelines). All patient with detectable viremia will be included, with selection of controls with viral suppression from the same cohort.

Approximately 800 newly diagnosed persons and 1600 ART recipients will be included (total estimated number of participants approximately 2400 individuals). Study investigations will be performed by project-employed research nurses. All eligible participants will receive oral and written information about the study. Tracing will be done by dedicated tracers. Study source data will be kept at the respective health facility. It will be coded and continuously recorded into a REDCAP database by project-employed staff.

Participants will be interviewed following structured questionnaires covering demographic, socio-economic, behavioral and medical details, as well as details on HIV testing and ART. For patients with prior and/or current HIV care history, previous VL and CD4 cell test results will be retrieved. Physical examination will be performed. Individuals with symptoms and/or signs of acute or chronic disease will be further investigated, depending on clinical presentation. Decisions on ART regimen will be done following Ethiopian guidelines.

Venous blood samples will be obtained in connection to inclusion, for VL, CD4 cell and complete blood count, serology for syphilis, hepatitis B and C. In addition, sputum samples will be obtained from all participants (irrespective of clinical manifestations) for bacteriological testing for Mycobacterium tuberculosis (including liquid culture and GeneXpert PCR). Stool samples will be analyzed microscopically for detection of intestinal worms and parasites. Investigation for other opportunistic infections will be performed depending on clinical presentation. Aliquots of plasma will be stored at -80° C.

Participants will be followed for 2 years after inclusion, with study visits at 3-monthly intervals during the first year and at 6-monthly intervals during the second year. On all visits, participants will be interviewed and examined, with repeated blood sampling for VL and CD4 cell count testing and storage of plasma as described above.

Analyses For characterization of HIV transmission patterns, data from phylogenetic analyses of viral sequences will be correlated to presence of drug-resistance mutations and socio-demographic characteristics. Samples with detectable VL (>150 copies/ml) will be subjected to PCR amplification of the entire protease-polymerase region (containing the three major regions associated with drug resistance; the protease, polymerase and integrase regions), followed by sequencing using 3rd generation sequencing technology. These sequences will be used for phylogenetic analysis, and for determination of HIV subtype, recombinant forms and presence of drug-resistance mutations. For further characterization of HIV transmission dynamics, avidity testing will be done on samples from newly diagnosed individuals, in order to estimate duration of HIV infection, and to identify persons with recently acquired HIV infection.

For analysis of treatment outcomes, participants will be followed for 2 years after inclusion. All samples with detectable VL obtained >3 months after inclusion will be subjected to sequencing for detection of drug-resistance mutations. Rates of viral suppression (defined as VL <150 copies/mL from 6 months after inclusion and onwards) will be compared between participant categories, with adjustment for co-variates potentially associated with these outcomes (sex, age, CD4 cell count, baseline VL, socio-demographic characteristics, presence of tuberculosis co-infection). Apart from virological outcomes, retention in care will be determined, with recording of mortality and loss to follow-up. In addition, analyses disaggregated by sex will be performed to detect sex-specific associations with treatment outcomes. For participants in whom drug-resistance mutations are detected at any time point, comparison with other sequences obtained from the same individual (including inclusion samples) will be done to assess longitudinal evolution of drug resistance. For this purpose, the presence of low frequencies of drug-resistance mutations (representing <1-2% of the viral population) will be determined separately.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent Positive HIV test result

Exclusion Criteria:

-

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People with HIV. Two categories of participants will be included: 1) persons with no prior or current exposure to antiretroviral therapy; 2) persons with prior or current exposure to antiretroviral therapy. From the latter group, all persons with detectable viremia will be included, with a similar total number of persons with viral suppression (and with no previous recorded lack of viral suppression during antiretroviral therapy).
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Clustering of HIV genomic sequences | 2023-2024
  Clustering indicating transmission between persons on antiretroviral therapy with lack of viral suppression and persons newly diagnosed with HIV

SECONDARY OUTCOMES:
Clustering of HIV genomic sequences with drug-resistance mutations | 2023-2024
  Clustering indicating transmission of viruses carrying drug-resistance mutations between persons on antiretroviral therapy with lack of viral suppression and persons newly diagnosed with HIV
Lack of viral suppression longitudinally during antiretroviral therapy | 2024-2026
  Viral load will be measured at defined time points during 2-year follow-up; levels above the detection limit (150 copies/ml) will define this outcome
Emergence of drug-resistance mutations longitudinally during antiretroviral therapy | 2024-2026
  Viremic samples (obtained at any time point during 2-year follow-up) will be sequenced for analysis of mutations associated with drug-resistance

CONTACTS AND LOCATIONS:
Overall Officials: Per Björkman, MD, PhD, Principal Investigator — Lund University; Alemseged Abdissa, PhD, Study Director — Armauer Hansen Research Institute
Locations (1):
- Public hospitals and health centers in the Adama uptake area, Ādama, Oromiya, Ethiopia

IPD SHARING:
Plan to Share IPD: Undecided